CLINICAL TRIAL: NCT01645891
Title: TCO2-2012-01 A Prospective, Randomized, Double-Blind Multicenter Study Comparing Continuous Diffusion of Oxygen (CDO) Therapy to Standard Moist Wound Therapy (MWT) in the Treatment of Diabetic Foot Ulcers
Brief Title: A Prospective, Randomized, Double-Blind Multicenter Study Comparing CDO Therapy to Standard MWT in the Treatment of DFUs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Electrochemical Oxygen Concepts, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TC02-2012-01
Record Dates: First submitted 2012-07-18; First posted 2012-07-20 (Estimated); Results first posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-09

CONDITIONS: Diabetic Foot Ulcer
Keywords: Diabetic Foot Ulcer
MeSH Terms: conditions — Diabetic Foot

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- CDO with standard MWT (Active Comparator): CDO (continuously supply pure oxygen) with standard Moist Wound Therapy
  Interventions: Device: CDO electrochemical tissue oxygenation system
- Moist Wound Therapy (Sham Comparator): Moist Wound Therapy. De-activated Sham device placed to wound in order to blind patient and study staff.
  Interventions: Device: Moist Wound Therapy

INTERVENTIONS:
Device: CDO electrochemical tissue oxygenation system — The TransCu O2® device is a non-invasive, electrochemical tissue oxygenation system intended for use with lower-cost wound dressings for the treatment of chronic wounds such as diabetic foot ulcers, venous leg ulcers, pressure ulcers and other skin wounds through the continuous diffusion of oxygen (CDO). The goal of CDO therapy is to continuously supply pure oxygen to an oxygen-compromised wound to aid in wound healing
  Other Names: TransCu O2® device; CDO Therapy
  Arms: CDO with standard MWT
Device: Moist Wound Therapy — Moist Wound Therapy in combination with sham or deactivated device
  Arms: Moist Wound Therapy

SUMMARY:
The purpose of this study was to evaluate the safety and effectiveness of Continuous Diffusion of Oxygen (CDO) therapy for the treatment of Diabetic Foot Ulcers. The primary objective of this study is to evaluate the effectiveness of CDO in combination with standard moist wound therapy (MWT) on wound healing as compared to standard MWT alone.

DETAILED DESCRIPTION:
This study was a 12-week, randomized, fully blinded, placebo-controlled, parallel group clinical trial evaluating the use of the CDO device for DFUs. The CDO device used was the TransCu O2 System. The study was approved by the Schulman Associates Institutional Review Board (Cincinnati, OH, IRB No. 201202439). Randomisation lists were made by the statistician for each clinical site in blocks of size four with SAS. Devices were labelled by the statistician before shipping to the sites. The sites assigned devices to patients sequentially at randomisation. Both arms received identical treatment (device, dressings, etc.) and the devices were functional in both arms with the exception that the oxygen did not flow to the ulcer in the placebo arm. All devices were functional in that they produced oxygen and displayed the oxygen flow rate. This had the effect that the devices appeared identical, including battery drain and oxygen flow display. The only difference was that the placebo devices did not have any oxygen flowing out of the oxygen supply port. Since the oxygen flow rate (3ml/ hour) is low enough that it cannot be felt by the subjects or physicians, the devices all appeared identical. Similarly, the dressings and offloading boots in each arm were limited and identical. The result was that the patients, doctors, evaluators, sponsor and statistician were all fully-blinded to the treatment arms until the data had been collected and verified, thereby eliminating the placebo effect.

Before assignment of a device, all patients were subjected to a run-in period during which they received standard of care dressings, debridement and off-loading to ensure that the wounds were indeed chronic in nature. There were two inclusion criteria essential to the design of the study to ensure that only chronic wounds were being included: initial or baseline wound size and initial or run-in rate of wound closure. These were defined as: 1) baseline DFU size: the ulcer area as determined by independently-verified digital planimetric analysis during screening through the randomization visit, and 2) run-in ulcer closure rate: the percentage of ulcer closure (percentage wound area reduction, or PWAR) during the run-in period before the placement of the device. All subjects received MWT during the run-in period.

The intent was to find a balance between a short run-in period and robust screening criteria to help ensure that non-chronic wounds were not included in the study. Since the PWAR assessment relied on independently-verified planimetric analysis of wound photos, some subjects were initially placed on a device at the conclusion of the run-in period and subsequently found to be not eligible for failing study inclusion/ exclusion criteria. These subjects were removed as not eligible.

The primary efficacy outcome was complete wound closure, defined as complete re-epithelialization with no drainage as assessed by the treating clinician and confirmed by a blinded observer.

ELIGIBILITY:
Inclusion Criteria:

* Subjects 30-90 years of age at the time of Informed Consent
* Subjects with type 1 or type 2 Diabetes Mellitus with a non-healing, full-thickness, University of Texas Classification of Diabetic Foot Ulcers Class IA diabetic foot ulcers
* Subjects who have an ulcer with a duration of at least 4 weeks, but not greater than 52 weeks at time of screening
* Subjects with an index ulcer measuring between 1.5 - 10 cm2 in area after debridement (Area = length x width) at time of Screening 1 and Screening 2, as measured using digital photography & computerized planimetric analysis by Centralized Wound Measuring Center (CWMC)
* Subjects with a diabetic foot ulcer(s) at or below the malleoli
* Subjects who demonstrates adequate arterial perfusion defined as either:

  * transcutaneous oxygen measurements of the dorsum of the foot > 30 mm Hg with a skin perfusion pressure > 30 mm Hg, or an ankle/brachial index (ABI) above 0.7, with documented confirmation of adequate arterial perfusion, or
  * a Doppler waveform consistent with adequate flow in the foot (biphasic or triphasic waveforms) at screening, or
  * absolute toe pressure of > 30 mm Hg
* Subject and/or caregiver must be able and willing to learn and perform the duties of dressing changes
* Subjects are able and willing to comply with standardized off-loading regimen (such as a fixed ankle walker)

Exclusion Criteria:

* Subjects < 30 or > 90 years of age at the time of Informed Consent

  * Subjects with Target Ulcers with a duration < 4 weeks or > 52 weeks
  * Subjects with ulcers measuring less than 1.5 cm2 or greater than 10 cm2 in area (Area = length x width) after debridement at the time of Screening 1 and Screening 2 to Randomization) or > 50% during the 2 week screening period, as measured using digital photography & computerized planimetric analysis's determined by CWMC.
  * Subjects whose ulcer decreased in area by > 30 % during the 1 week screening period
  * Subjects with evidence of gangrene on any part of affected limb
  * Subjects with active Charcot's foot on the study limb
  * Subjects scheduled to undergo vascular surgery, angioplasty or thrombolysis at the time of enrollment
  * Subjects with active infection at the time of screening
  * Subjects with a target ulcer which has exposed tendons, ligaments, muscle, or bone
  * Subjects with active malignancy, excluding non-melanoma skin cancer
  * Subjects with a history of malignancy on study limb
  * Subjects in whom oral, or IV antibiotic/antimicrobial agents or medications have been used within 2 days (48 hours) of baseline
  * Subjects who are currently receiving or has received radiation or chemotherapy within 3 months of randomization
  * Subjects who have received growth factor therapy (e.g., autologous platelet-rich plasma gel, becaplermin, bilayered cell therapy, dermal substitute, extracellular matrix) within two weeks of screening
  * Subjects who are pregnant at the time of screening
  * Subjects who are undergoing active renal dialysis
  * Subjects who have a known immune insufficiency, excluding Diabetes Mellitus
  * Subjects with a history of peripheral vascular repair within 14 days of screening
  * Subjects with a current deep vein thrombosis (DVT)
  * Subjects with ulcers due to Raynaud's disease
  * Subjects with and ulcer due to acute thrombophlebitis
  * Subjects with inadequate perfusion to support healing
  * Subjects with necrotic wounds covered with eschar or slough
  * Subjects with wounds with fistulae or deep sinus tracts of unknown depth
  * Subjects who are receiving palliative care
  * Subjects who have a HbA1c > 12% (uncontrolled hyperglycemia)
  * Subjects whose target ulcer has a known etiology of: malignancy, burn, collagen vascular disease, sickle cell, vasculopathy, or pyoderma gangrenosum
  * Subjects with a documented history of alcohol or substance abuse within 6 months of screening
  * Subjects who are currently enrolled or who have participated, within 30 days of screening, in another investigational device, drug or biological trial that may interfere with study results
  * Subjects with a known allergy to dressing materials, including occlusive dressings and the adhesives on such dressings

Ages: 30 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 146 (Actual)
Dates: Start 2012-04; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David G Armstrong, DPM, MD, PhD, Principal Investigator — Southern Arizona Limb Salvage Alliance (SALSA)
Locations (33):
- United States (33):
  - Clinical Trials of Texas, Inc., dba Clinical Trials of Arizona, Inc., Glendale, Arizona
  - Associated Foot and Ankle Specialists, Phoenix, Arizona
  - Premier Foot & Ankle Surgeons, Tucson, Arizona
  - Southern Arizona VA Health Care System, Tucson, Arizona
  - Sacramento Foot & Ankle Center, Fair Oaks, California
  - Roy O. Kroeker, DPM , Inc., Fresno, California
  - Limb Preservation Platform, Fresno, California
  - Center for Clinical Research, Inc, San Francisco, California
  - The Research Center, Hialeah, Florida
  - Phoenix Medical Research, Miami, Florida
  - Doctors Research Network, South Miami, Florida
  - Orthopedic Research Institute, West Palm Beach, Florida
  - Aiyan Diabetes Center, Martinez, Georgia
  - Weil Foot & Ankle Institute, Chicago, Illinois
  - Weil Foot & Ankle Institute, Des Plaines, Illinois
  - Foot and Ankle Specialists of the Mid-Atlantic, Annapolis, Maryland
  - Foot and Ankle Specialists of the Mid-Atlantic, Kensington, Maryland
  - Foot and Ankle Specialists of the Mid-Atlantic, Pasadena, Maryland
  - Clinical Research Medical Center, Las Vegas, Nevada
  - Impact Clinical Trials, Las Vegas, Nevada
  - PMG Research of Salisbury, Salisbury, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Clinical Research Associates of Central PA, Altoona, Pennsylvania
  - Foot and Ankle Center, Haverford, Pennsylvania
  - Integrated Clinical Research, Abilene, Texas
  - Richard C. Galperin, DPM, PA, Dallas, Texas
  - William Blake Partners, LLC, Grapevine, Texas
  - Houston Foot & Ankle, Houston, Texas
  - Complete Family Foot Care, McAllen, Texas
  - Alamo Clinical Research, San Antonio, Texas
  - Clinical Trials of Texas, San Antonio, Texas
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Clinical Research Medical Center, Salt Lake City, Utah

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Patients were monitored for 2 weeks with SOC prior to randomization. Subjects with wounds that failed inclusion/exclusion criteria or closed too quickly (non-chronic) via planimetric analysis were excluded or removed from the study. Of 386 screened patients, 146 met inclusion criteria and participated in the treatment phase.
Groups:
- Active Arm - Moist Wound Therapy With Active CDO Device: CDO (Continuous Diffusion of Oxygen) with standard Moist Wound Therapy. CDO electrochemical tissue oxygenation system: The TransCu O2® device is a non-invasive, electrochemical tissue oxygenation system intended for use with lower-cost wound dressings for the treatment of chronic wounds such as diabetic foot ulcers, venous leg ulcers, pressure ulcers and other skin wounds through the CDO. The goal of CDO therapy is to continuously supply pure oxygen to an oxygen-compromised wound to aid in wound healing. The active arm is basically moist wound therapy plus a continuous infusion of pure, humidified oxygen. Dressings, offloading and standard of care are identical in both arms.
- Placebo Arm - Moist Wound Therapy With Sham CDO Device: Moist Wound Therapy with Sham CDO Device. A fully functional sham device is used in order to blind patient and study staff. The sham device is functional, producing oxygen and identical to active device with the exception that the oxygen diverted within the device and no oxygen was delivered to the wound bed. Thus, the placebo arm appears identical to the the active arm with the goal of achieving full study blinding. Dressings, offloading and standard of care are identical in both arms.
Period: Overall Study
Arm/Group | Active Arm - Moist Wound Therapy With Active CDO Device | Placebo Arm - Moist Wound Therapy With Sham CDO Device
Started | 74 | 72
Completed | 52 | 53
Not Completed | 22 | 19
Not completed — Adverse Event | 6 | 10
Not completed — Adverse Event Unrelated to Wound | 5 | 3
Not completed — Withdrawal by Subject | 3 | 3
Not completed — Protocol Violation | 4 | 0
Not completed — Lost to Follow-up | 4 | 1
Not completed — Death | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active Arm - Moist Wound Therapy With Active CDO Device | Placebo Arm - Moist Wound Therapy With Sham CDO Device | Total
Number analyzed (Participants) | 74 | 72 | 146
Age, Continuous [Mean (Standard Deviation); unit: Years] | 56.1 (10.1) | 56.6 (14.4) | 56.3 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15 | 18 | 33
  Male | 59 | 54 | 113
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 29 | 55
  Not Hispanic or Latino | 47 | 43 | 90
  Unknown or Not Reported | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 12 | 25
  White | 60 | 60 | 120
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 74 | 72 | 146
Wound Area, cm^2 ± SD [Mean (Standard Deviation); unit: cm^2] | 3.54 (1.68) | 3.89 (2.02) | 3.71 (1.85)
Wound Age, days ± SD [Mean (Standard Deviation); unit: years] | 131.6 (89.2) | 143.8 (97.7) | 137.6 (93.4)
Hemoglobin A1C (HbA1c) ± SD [Mean (Standard Deviation); unit: %] | 8.4 (1.6) | 8.3 (2) | 8.3 (1.8)
Ankle Brachial Index (ABI) ± SD [Mean (Standard Deviation); unit: index units] — The purpose of the ABI is to support the diagnosis of vascular disease by providing an objective indicator of arterial perfusion to a lower extremity. ABI is performed using a continuous wave Doppler, a sphygmomanometer and pressure cuffs to measure brachial and ankle systolic pressures. ABI is a ratio derived from dividing the higher of the ankle pressures for each leg by the higher of the right and left arm's brachial systolic pressures. An ABI of 0.9 or higher is considered normal, with higher numbers being better, whereas an ABI of 0.9 or lower indicates compromised blood flow.
  index units | 1.05 (.14) | 1.02 (.15) | 1.03 (.15)
Participants with Wound Weight Bearing Surface [Number; unit: participants] | 59 | 53 | 112
Participants with No Wound Pain at Baseline [Count of Participants; unit: Participants] — This measure depicts whether the participant had a pain score of zero (0) "No Wound Pain" on a scale of 0-10 at the baseline visit. Any values from 1-10 were registered as "Wound Pain" Population: This measure depicts whether the participant had a pain score of zero (0) on a scale of 0-10 at the baseline visit. There was one participant in each arm (2 total) for which a baseline pain score was not recorded. Therefore the total number of participants with pain scores does not match the total number of participants: the total with pain scores at baseline is 144 whereas the total number of participants is 146.
  Participants
    number analyzed (Participants) | 73 | 71 | 144
    (all) | 32 | 26 | 58
Participants with Wound Pain at Baseline [Count of Participants; unit: Participants] — This measure depicts whether the participant had a pain score of zero (0) "No Wound Pain" on a scale of 0-10 at the baseline visit. Any values from 1-10 were registered as "Wound Pain". Population: There was one participant in each arm (2 total) for which a baseline pain score was not recorded. Therefore the total number of participants with pain scores does not match the total number of participants: the total with pain scores at baseline is 144 whereas the total number of participants is 146.
  Participants
    number analyzed (Participants) | 73 | 71 | 144
    (all) | 41 | 45 | 86

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete (100%) Wound Closure Defined as Complete Re-epithelialization Without Drainage
Description: Number of Participants with complete (100%) wound closure defined as complete re-epithelialization without drainage before or at week 12
Time Frame: 12 weeks or wound closure
Population: Subjects who completed the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Active Arm - Moist Wound Therapy With Active CDO Device | Placebo Arm - Moist Wound Therapy With Sham CDO Device
Number analyzed (Participants) | 52 | 53
Participants | 24 | 12

2. Secondary Outcome: Time to 50% Wound Closure
Description: Time to 50% wound closure by using digital photography & computerized planimetric analysis
Time Frame: 12 weeks or wound closure
Population: All eligible patients, including patients who dropped from the study, were analyzed for time (in days) to reach 50%, 75% and 100% wound closure via planimetric analysis.
Measure: Median (Standard Deviation); unit: days
Arm/Group | Active Arm - Moist Wound Therapy With Active CDO Device | Placebo Arm - Moist Wound Therapy With Sham CDO Device
Number analyzed (Participants) | 74 | 72
days | 18.45 (16.32) | 28.9 (22.54)

3. Secondary Outcome: Time to 75% Wound Closure
Description: Time to 75% wound closure by using digital photography & computerized planimetric analysis
Time Frame: 12 weeks or wound closure
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: days
Arm/Group | Active Arm - Moist Wound Therapy With Active CDO Device | Placebo Arm - Moist Wound Therapy With Sham CDO Device
Number analyzed (Participants) | 74 | 72
days | 27.8 (19.89) | 40 (15.46)

4. Secondary Outcome: Time to 100% Wound Closure
Description: Time to 100% wound closure by using digital photography & computerized planimetric analysis
Time Frame: 12 weeks or wound closure
Population: as for outcome 2
Measure: Median (Standard Deviation); unit: days
Arm/Group | Active Arm - Moist Wound Therapy With Active CDO Device | Placebo Arm - Moist Wound Therapy With Sham CDO Device
Number analyzed (Participants) | 74 | 72
days | 49 (18.17) | 59.5 (21.22)

ADVERSE EVENTS:
Time Frame: 24 weeks
Arm/Group | Active Arm - Moist Wound Therapy With Active CDO Device | Placebo Arm - Moist Wound Therapy With Sham CDO Device
All-Cause Mortality (participants affected / at risk) | 0/74 | 2/72
Serious Adverse Events (participants affected / at risk) | 0/74 | 0/72
Other Adverse Events (participants affected / at risk) | 11/74 | 13/72
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active Arm - Moist Wound Therapy With Active CDO Device (N=74) | Placebo Arm - Moist Wound Therapy With Sham CDO Device (N=72)
Infection (Skin and subcutaneous tissue disorders) | 6 (6) | 10 (10) — Infections related to study wound of interest. Two infections in Placebo Arm had Gangrene, zero in the Active Arm
Traffic accident (Social circumstances) | 1 (1) | 0 (0) — Patient involved in traffic accident leaving study site, unrelated to study wound or treatment
Osteomyelitis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — Subject experienced osteomyelitis in wound other than study wound, unrelated to study wound or treatment
New Abcess (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) — New wound formed, unrelated to study wound or treatment
Anemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) — Unrelated to study wound or device
Drug Overdose (Social circumstances) | 0 (0) | 1 (1) — Drug overdose and potential suicide, unrelated to study wound or treatment
Infection, Abscess, Cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — Unrelated wound, study wound not affected, unrelated to study wound or treatment
Arterial Stenosis (Blood and lymphatic system disorders) | 2 (2) | 0 (0) — Femoral Arterial Stenosis unrelated to study wound or treatment

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No